CLINICAL TRIAL: NCT04006600
Title: Is There a Link Between Anatomical Markers of Surgical Difficulty and Incapacity to Reverse Stoma After Low Rectal Cancer Surgery?
Acronym: persist stomie
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local 2018/MB-02
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Rectal Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sphincter saving proctectomy — After rectal resection, when colorectal anastomosis is subperitoneal, it is currently recommended to perform a protective stoma to reduce the potential consequences of a fistula. This stoma, which is intended to be temporary, appears to be permanent in 6 to 32% of cases in the literature.
  The objective of the study is therefore to look for a statistical link between the persistence of a permanent stoma and the intraoperative difficulty represented by pelvic anatomical stress.

SUMMARY:
Anterior resection with total mesorectal excision (TME) is the standard procedure for mid and low rectal cancers . A colo-rectal anastomosis under peritoneal reflection is, most of the time, protected by a temporary loop stoma to decrease the risk and severity of anastomotic morbidity. This stoma, which is intended to be temporary, appears to be permanent in 6 to 32% of cases in the literature. The main risk factor being anastomotic leakage. Two major risk factors for anastomotic leakage after colorectal surgery are " male sex " and " Body mass index ", which are responsible of a higher anatomical difficulty (Narrow pelvis and bulky mesorectal fat) Therefore, the objective of this study is to look for a statistical link between permanent stoma and intraoperative difficulty represented by pelvic anatomical constraints.

DETAILED DESCRIPTION:
Anterior resection with total mesorectal excision (TME) is the standard procedure for mid and low rectal cancers . A colo-rectal anastomosis under peritoneal reflection is, most of the time, protected by a temporary loop stoma to decrease the risk and severity of anastomotic morbidity. This stoma, which is intended to be temporary, appears to be permanent in 6 to 32% of cases in the literature. The main risk factor being anastomotic leakage. Two major risk factors for anastomotic leakage after colorectal surgery are " male sex " and " Body mass index ", which are responsible of a higher anatomical difficulty (Narrow pelvis and bulky mesorectal fat) Studies focused on surgical difficulties usually evaluated criteria such as, total surgery duration, blood loss or surgeon's subjective evaluation. The investigators of this retrospective study hypothesize that when a stoma,primarily intended to be temporary, is not reversed after a long (2 years) post operative delay, it all comes to surgical difficulties and that these surgical difficulties are essentially represented by anatomical constraints. Therefore, the objective of this study is to look for a statistical link between permanent stoma and intraoperative difficulty represented by pelvic anatomical constraints.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent a sphincter saving resection for low rectal cancer between January 2019 and December 2017.

Exclusion Criteria:

* Minor patients.
* Patients who have undergone a cancer proctectomy with no restoration of continuity expected.
* Patients who did not have total Mesorectal excision

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent a cancer proctectomy with sphincter conservation
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Persistence of a stomy 2 years after rectal surgery when stoma was primarily intended to be temporary | 2 years
  Number of patient with the persistence of a permanent stoma

CONTACTS AND LOCATIONS:
Overall Officials: Martin BERTRAND, Principal Investigator — Nîmes University Hospital
Locations (1):
- Nimes University Hospital, Nîmes, France